CLINICAL TRIAL: NCT03005483
Title: Placebo Controlled, Randomized,Gabapentin as Adjuvant for Postoperative Pain in Pediatric Orthopedic Surgery
Brief Title: Gabapentin as Adjuvant for Postoperative Pain in Pediatric Orthopedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Infantil Albert Sabin (Other)
Collaborators: Fortaleza University (Other)
Responsible Party: Principal Investigator, washington aspilicueta pinto filho, Medical Anesthesiologist, Hospital Infantil Albert Sabin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOSPITALIAS
Record Dates: First submitted 2016-12-13; First posted 2016-12-29 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Pain, Postoperative; Orthopedic Disorder
Keywords: GABAPENTIN POSTOPERATIVE PAIN CHILD
MeSH Terms: conditions — Pain, Postoperative; Musculoskeletal Diseases | interventions — Gabapentin; Orthopedic Procedures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): Gabapentin 10 mg/kg in children submitted unilateral limb surgery
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Placebo in children submitted unilateral limb surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Orthopedic Surgery was applied for the treatment of osseous disorders
  Other Names: Orthopedic Surgery
  Arms: Gabapentin
Other: Placebo — Orthopedic Surgery was applied for the treatment of osseous disorders
  Arms: Placebo

SUMMARY:
This study is a clinical trial, prospective, randomized and double-blinded. Gabapentin oral 10 mg/kg was administered to reduce the pain intensity as well as the opioid consumption in children from 3 months to 16 years submitted unilateral limb surgery.

DETAILED DESCRIPTION:
This study is a clinical trial, prospective, randomized and double-blinded. Gabapentin oral 10 mg/kg was administered to reduce the pain intensity as well as the opioid consumption in children from 3 months to 16 years submitted unilateral limb surgery. The children were divided into 2 groups: the gabapentin group (GG) was administered gabapentin 1 to 2 hours before procedure (N-40) and the placebo group (GP) was administered placebo 1 to 2 hours before surgery (N-44). Both groups were subjected to the same general anesthesia protocol, opioid free, and femoral and sciatic block with bupivacaine 0.125%. All patients received dipyrone and rescue analgesic used was morphine into 2/2h. The variables studied were age, gender, weight, type of surgery, hemodynamics, postoperative pain and morphine consumption .

ELIGIBILITY:
Inclusion Criteria:

Children between 3 months and 16 years who were previously healthy submitted to unilateral lower limb surgery

Exclusion Criteria:

Children cardiac, pulmonary, renal and neurological diseases and allergy and refusal of parents, caregivers and patients to participate in the study.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduce the pain intensity using the Face Pain Scale | 24 hour
  Subjected to the same general anesthesia protocol, opioid free, and femoral and sciatic block with bupivacaine 0.125%.The evaluation times were: 1 hour, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours after surgery. The time elapsed was recorded, from the end of the surgery to the first use of morphine. The parents and the patients themselves were instructed to request analgesic at any time.

SECONDARY OUTCOMES:
Reduce the opioid consumption through 24 hours postoperative observation | 24 hour
  Subjected to the same general anesthesia protocol, opioid free, and femoral and sciatic block with bupivacaine 0.125%. All patients received dipyrone and rescue analgesic used was administered morphine 50mcg / kg (maximum dose of 2mg) up to 2 / 2h when Face´s Scales reached 5 points.

CONTACTS AND LOCATIONS:
Overall Officials: Josenília Gomes, PhD, Study Chair — Fortaleza University
Locations (1):
- Hospital Infantil Albert Sabin, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rusy LM, Hainsworth KR, Nelson TJ, Czarnecki ML, Tassone JC, Thometz JG, Lyon RM, Berens RJ, Weisman SJ. Gabapentin use in pediatric spinal fusion patients: a randomized, double-blind, controlled trial. Anesth Analg. 2010 May 1;110(5):1393-8. doi: 10.1213/ANE.0b013e3181d41dc2. PMID 20418301
- [Background] Mayell A, Srinivasan I, Campbell F, Peliowski A. Analgesic effects of gabapentin after scoliosis surgery in children: a randomized controlled trial. Paediatr Anaesth. 2014 Dec;24(12):1239-44. doi: 10.1111/pan.12524. Epub 2014 Sep 17. PMID 25230144